CLINICAL TRIAL: NCT03893695
Title: Combination of GT90001 and Nivolumab in Patients With Metastatic Hepatocellular Carcinoma
Brief Title: Combination of GT90001 and Nivolumab in Patients With Metastatic Hepatocellular Carcinoma(HCC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Kintor Pharmaceutical Inc, (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GT90001-TW-1001
Record Dates: First submitted 2019-03-21; First posted 2019-03-28 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Hepatocellular Carcinoma; HCC; Combinations of Drugs; Dependence
Keywords: Phase Ib/II; HCC; Metastatic Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Single arm, Open label,Two stage study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- metastatic HCC (Experimental): Stage one - Dose de-escalation:
  Each dose cohort will assess toxicity within the 28 days following the first dose of nivolumab and GT90001.
  Stage two- the expansion cohort:
  14 patients will be enrolled to the expansion cohort where one or no DLT takes place in planned study cohort.
  Interventions: Drug: GT90001 and Nivolumab

INTERVENTIONS:
Drug: GT90001 and Nivolumab — Stage1:Dose de-escalation. Stage2:the expansion cohort where one or no DLT takes place in planned study cohort.
  Other Names: GT90001 and Opdivo

SUMMARY:
This single arm, open label, two stage study will be conducted in several medical centers around Taiwan. Stage one determine safety and tolerability in patients with HCC, and stage two assess anti-tumor activities of GT90001 in combination with nivolumab in patients with metastatic HCC. Subjects who fulfill all the entry criteria and have written informed consent will be enrolled to the study.

DETAILED DESCRIPTION:
Based on published and first-hand experience with the safety and tolerability of both GT90001 and nivolumab, the proposed dose is GT90001 7 mg/kg in combination with nivolumb 3 mg/kg. Nivolumab will first be administered by intravenous infusion over 60 minutes, then 30 minutes later, give GT90001 intravenous infusion for 1 hour. All participants will receive GT90001 + Nivolumab until unacceptable toxicity, disease progression or loss of clinical benefit as determined by the investigator.The primary objective of the study is to determine the safety and tolerability of GT90001 in combination with nivolumab in subjects with advanced and or metastatic HCC who were progressed on or were intolerant of first-line and/or second-line systemic therapy. The secondary objectives will be to evaluate the anti-tumor efficacy and the PK profile of this combination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial;
2. Age ≥20 years male and female;
3. Subjects must have confirmed diagnosis of unresectable HCC with any of following criteria:

   i. Histologically or cytologically confirmed diagnosis of HCC ii. Have Barcelona Clinic Liver Cancer (BCLC) Stage C disease or BCLC Stage B disease not amenable to locoregional therapy or refractory to locoregional therapy;
4. Have documented disease progression or intolerance after first-line systemic treatment;
5. At least one measurable lesion based on RECIST version 1.1 ;
6. Child-Pugh score ≤ 6 (Child-Pugh A)score within 7 days of first dose of study drug;
7. ECOG performance status: 0-1;
8. Have a predicted life expectancy of greater than 3 months;
9. The functions of the important organs are confirmed with the following requirement:

   * Hemoglobin (HGB) ≥ 90 g/L;
   * White blood cell count (WBC) ≥ 3×10^9/L；
   * Absolute neutrophil count (ANC) ≥ 1.5×10^9/L；
   * Platelets (PLT) ≥ 100×10^9/L；
   * Total bilirubin (TBIL) ≤ 1.5× Upper limit of normal value (ULN)
   * Aspartate aminotransferase (AST), alkaline phosphatase (ALP), and alanine aminotransferase (ALT) ≤ 5× ULN
   * Creatinine (Cr) ≤ 1.5×ULN；
   * International normalization ratio (INR)or prothrombin time (PT) ≤ 1.5×ULN ;
10. Women must have a negative serum or urine pregnancy test within 72 hours prior to the start of investigational product;
11. Women of childbearing potential must agree to contraception for the duration of study treatment and 5 months after the last dose of study treatment;
12. Willing and able to comply with all aspects of the protocol

Exclusion Criteria:

1. Imaging findings for HCC corresponding to any of the following:

   * HCC with ≥ 50% liver occupation
   * Clear invasion into the bile duct
   * Portal vein invasion or thrombosis at the main portal branch (Vp4)
2. Gastric or esophageal varices that require treatment;
3. If prior history of DVT/PE, the patient needs to be on stable doses of anticoagulation with low molecular weight heparin or oral anticoagulant for at least two weeks;
4. Esophageal vein dilation, grade A of active peptic ulcer rating, and all bleeding risk by gastroscopy;
5. History of arterial thromboembolic event in past 6 months;
6. Active bleeding disorder, including gastrointestinal bleeding event or active hemoptysis within 28 days prior to study treatment;
7. Have central nervous system (CNS) metastases;
8. Has a known history of human immunodeficiency virus (HIV);
9. Has received prior immune checkpoint inhibitor (including those targeting PD-1, PD-L1 or PD-L2, CD137, or cytotoxic T-lymphocyte antigen [CTLA-4]);
10. Has a known history of, or any evidence of, interstitial lung disease or active non- infectious pneumonitis;
11. Has active autoimmune disease that has required systemic treatment in past 2 years;
12. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial;
13. Any history of drug or alcohol dependency or abuse within the prior 1 years;
14. Has known active Hepatitis B or Hepatitis C within 2 weeks prior to initiation of study treatment Note: Patients with HBV infection are required to be receiving effective antiviral therapy over two weeks, and then have continuous therapy in study period;
15. Pregnant, breast feeding, or planning to become pregnant;
16. Have a history of severe hypersensitivity reaction to monoclonal antibody;
17. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke within 6 months of the first dose of study drug;
18. Have surgery, radiotherapy, ablation within one month before screening;
19. Subjects with any other serious disease considered by the investigator not in the condition to enter into the trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-25 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
Dose-limiting Toxicity(DLT) | 28 days
  Each dose cohort will initially include 6 evaluable patients for assessment of toxicity within the 28 days following the first dose of nivolumab and GT90001.

SECONDARY OUTCOMES:
overall response rate (ORR) | 2 years
  To estimate ORR, per RECIST 1.1 assessed by investigator review
the duration of response (DOR), | 2 years
  To evaluate the DOR per RECIST 1.1 assessed by investigator review
disease control rate (DCR), | 2 years
  To evaluate the DCR per RECIST 1.1 assessed by investigator review
time to response (TTR) | 2 years
  To evaluate the TTR per RECIST 1.1 assessed by investigator review
progression-free survival (PFS) | 2 years
  To evaluate the PFS per RECIST 1.1 assessed by investigator review
maximum concentration (Cmax) | 2 years
  Pharmacokinetics
time that maximum concentration is observed (tmax) | 2 years
  Pharmacokinetics
area under the concentration time-curve from time zero to infinity (AUC0∞) | 2 years
  Pharmacokinetics
area under the plasma concentration-time curve from time zero hours to time (t hrs), (AUC0-t) | 2 years
  Pharmacokinetics
area under the plasma concentration-time curve from time zero hours to 24 hours (AUC0-24) | 2 years
  Pharmacokinetics
terminal elimination rate constant (λz) | 2 years
  Pharmacokinetics
terminal elimination half life (t½) | 2 years
  Pharmacokinetics
volume of distribution (Vz) | 2 years
  Pharmacokinetics
volume of plasma cleared of the drug per unit time (C) | 2 years
  Pharmacokinetics
Exploratory Biomarker: circulating tumor deoxyribonucleic acid (ctDNA) | 2 years
  HCC-related pathway alterations including VEGF and TGF-β pathway genes

CONTACTS AND LOCATIONS:
Overall Officials: Yuwei Xu, Study Director — Suzhou Kintor Pharmaceuticals,inc.
Locations (3):
- Taiwan (3):
  - National Cheng Kung University Hospital, Tainan
  - MacKay Memorial Hospital, Taipei
  - National TaiWan University Hospital, Taipei

REFERENCES:
- [Derived] Hsu C, Chang YF, Yen CJ, Xu YW, Dong M, Tong YZ. Combination of GT90001 and nivolumab in patients with advanced hepatocellular carcinoma: a multicenter, single-arm, phase 1b/2 study. BMC Med. 2023 Oct 20;21(1):395. doi: 10.1186/s12916-023-03098-w. PMID 37858184